CLINICAL TRIAL: NCT04286672
Title: Serum Metadherin mRNA Expression in Bladder Cancer
Brief Title: Metadherin mRNA Expression in Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Nasr Abd-el-hakim, Principal Investigator, Assiut University
Other Study IDs: MmBC
Record Dates: First submitted 2020-02-17; First posted 2020-02-27 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:: • 35 bladder cancer patients diagnosed by biopsy before treatment.
  Interventions: Diagnostic Test: Metadherin
- Group 2:: 35 apparently healthy individuals who were matched by age and sex .
  Interventions: Diagnostic Test: Metadherin

INTERVENTIONS:
Diagnostic Test: Metadherin — study alterations of MTDH gene expression in the serum of bladder cancer patients

SUMMARY:
The study aims to study alterations of MTDH gene expression in the serum of bladder cancer patients compared to control group to evaluate its role as a marker for diagnosis.

,to compare the diagnostic accuracy of MTDH with the previously used marker Bladder Cancer-Specific Antigen-1 (BLCA-1 in the serum of bladder cancer patients .

and to study correlation between expression of the metadherin gene and serum level of BLCA-1, and clinical and histopathological staging in patients with bladder cancer

DETAILED DESCRIPTION:
Urinary bladder cancer (BC) is the ninth most common cancer worldwide. It is the fifth most common malignancy in males and seventeenth most common in females.

In Egypt, bladder cancer represents a massive health burden where it is one of the commonest cancers representing 6.9% in both sexes and 10.7% among men. Its distribution is 8.8% in lower Egypt, 14.2% in middle Egypt and 12.6% in upper Egypt.Almost 50% of patients will experience recurrence of their disease within 4 years of their initial diagnosis.The prognosis of bladder cancer is poor as a result of highly invasive properties of tumour cells.

The optimal treatment selection depends on early diagnosis as well as accurate staging and grading.Currently there is a need for new molecular bio markers that can help clinicians to identify patients requiring early, aggressive treatment.

Metadherin (MTDH) is an oncogene known as Astrocytic elevated gene-1(AEG-1).It was firstly identified in 2002 at fetal astrocytes of persons exposed to HIV-1 and then known as a vital oncogene mediating carcinogenesis,prognosis,invasion and cancer metastasis. AEG-1 expression is raised in bladder cancer tissues relative to normal tissues, and serves as a poor prognostic factor.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* 30-80 years old.
* patients with bladder cancer not receiving any treatment

Exclusion Criteria:

1. patients taking chemotherapy or radiotherapy.
2. History of other malignancy.
3. History of autoimmune diseases.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 1: 35 bladder cancer patients diagnosed by biopsy before treatment.
  * Group 2: 35 apparently healthy individuals who were matched by age and sex .
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
early diagnosis of bladder cancer patient | baseline
  study mRNA MTDH expression in the serum of bladder cancer patients compared to control group to evaluate its role as a marker for diagnosis.

SECONDARY OUTCOMES:
non invasive marker for detection of bladder cancer. | baseline
  To compare the diagnostic accuracy of MTDH with the previously used marker Bladder Cancer-Specific Antigen-1 (BLCA-1 in the serum of bladder cancer patients .

CONTACTS AND LOCATIONS:
Overall Officials: Lubna M. Tag El-Din, Doctorate, Study Chair — Lubna Mohamed Tag El-Din

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Rahman O, Helbling D, Schob O, Eltobgy M, Mohamed H, Schmidt J, Giryes A, Mehrabi A, Iype S, John H, Tekbas A, Zidan A, Oweira H. Cigarette smoking as a risk factor for the development of and mortality from hepatocellular carcinoma: An updated systematic review of 81 epidemiological studies. J Evid Based Med. 2017 Nov;10(4):245-254. doi: 10.1111/jebm.12270. Epub 2017 Sep 10. PMID 28891275
- [Result] Burger M, Catto JW, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol. 2013 Feb;63(2):234-41. doi: 10.1016/j.eururo.2012.07.033. Epub 2012 Jul 25. PMID 22877502
- [Result] Giopanou I, Bravou V, Papanastasopoulos P, Lilis I, Aroukatos P, Papachristou D, Kounelis S, Papadaki H. Metadherin, p50, and p65 expression in epithelial ovarian neoplasms: an immunohistochemical study. Biomed Res Int. 2014;2014:178410. doi: 10.1155/2014/178410. Epub 2014 May 22. PMID 24963474
- [Result] Guszcz T, Szymanska B, Kozlowski R, Lukaszewski Z, Laskowski P, Gorodkiewicz E. Plasma aromatase as a sensitive and selective potential biomarker of bladder cancer and its role in tumorigenesis. Oncol Lett. 2020 Jan;19(1):562-568. doi: 10.3892/ol.2019.11080. Epub 2019 Nov 11. PMID 31897172
- [Result] Hu B, Emdad L, Kegelman TP, Shen XN, Das SK, Sarkar D, Fisher PB. Astrocyte Elevated Gene-1 Regulates beta-Catenin Signaling to Maintain Glioma Stem-like Stemness and Self-Renewal. Mol Cancer Res. 2017 Feb;15(2):225-233. doi: 10.1158/1541-7786.MCR-16-0239. Epub 2016 Nov 30. PMID 27903708
- [Result] Kang DC, Su ZZ, Sarkar D, Emdad L, Volsky DJ, Fisher PB. Cloning and characterization of HIV-1-inducible astrocyte elevated gene-1, AEG-1. Gene. 2005 Jun 20;353(1):8-15. doi: 10.1016/j.gene.2005.04.006. PMID 15927426
- [Result] Li G, Wang Z, Ye J, Zhang X, Wu H, Peng J, Song W, Chen C, Cai S, He Y, Xu J. Uncontrolled inflammation induced by AEG-1 promotes gastric cancer and poor prognosis. Cancer Res. 2014 Oct 1;74(19):5541-52. doi: 10.1158/0008-5472.CAN-14-0968. Epub 2014 Aug 4. PMID 25092897
- [Result] Pan Y, Guo X, Yang Z, Chen S, Lei Y, Lin M, Wang L, Feng C, Ke Z. AEG-1 activates Wnt/PCP signaling to promote metastasis in tongue squamous cell carcinoma. Oncotarget. 2016 Jan 12;7(2):2093-104. doi: 10.18632/oncotarget.6573. PMID 26689985
- [Result] Park SY, Choi M, Park D, Jeong M, Ahn KS, Lee J, Fisher PB, Yun M, Lee SG. AEG-1 promotes mesenchymal transition through the activation of Rho GTPases in human glioblastoma cells. Oncol Rep. 2016 Nov;36(5):2641-2646. doi: 10.3892/or.2016.5106. Epub 2016 Sep 19. PMID 27667169
- [Result] Sarkar D, Park ES, Emdad L, Lee SG, Su ZZ, Fisher PB. Molecular basis of nuclear factor-kappaB activation by astrocyte elevated gene-1. Cancer Res. 2008 Mar 1;68(5):1478-84. doi: 10.1158/0008-5472.CAN-07-6164. PMID 18316612
- [Result] Su ZZ, Kang DC, Chen Y, Pekarskaya O, Chao W, Volsky DJ, Fisher PB. Identification and cloning of human astrocyte genes displaying elevated expression after infection with HIV-1 or exposure to HIV-1 envelope glycoprotein by rapid subtraction hybridization, RaSH. Oncogene. 2002 May 16;21(22):3592-602. doi: 10.1038/sj.onc.1205445. PMID 12032861
- [Result] Zhang L, Yang G, Chen H, Huang Y, Xue W, Bo J. Depletion of astrocyte elevated gene-1 suppresses tumorigenesis through inhibition of Akt activity in bladder cancer cells. Am J Transl Res. 2017 Dec 15;9(12):5422-5431. eCollection 2017. PMID 29312494